CLINICAL TRIAL: NCT01404117
Title: A Multinational, Randomized, Double-blind, Parallel-group, Placebo-controlled Study Assessing the Safety and Tolerability
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is being redesigned
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAQ-MS-201
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Laquinimod 0.6 (Experimental): GA 20 mg/1mL or an IFN-B preparation + oral daily administration of laquinimod 0.6 mg
  Interventions: Drug: Laquinimod 0.6
- Laquinimod 1.2 (Experimental): GA 20 mg/1mL or an IFN-B preparation + oral daily administration of laquinimod 1.2 mg
  Interventions: Drug: Laquinimod 1.2
- GA or IFN + Placebo (Experimental): GA 20 mg/1mL or an IFN-B preparation + oral daily placebo
  Interventions: Other: Glatiramer Acetate or interferon-beta+ Placebo

INTERVENTIONS:
Drug: Laquinimod 0.6 — Laquinimod 0.6 capsule
  Arms: Laquinimod 0.6
Drug: Laquinimod 1.2 — Placebo
  Arms: Laquinimod 1.2
Other: Glatiramer Acetate or interferon-beta+ Placebo — GA 20 mg/1mL or IFN-B (Avonex®, Betaseron®/Betaferon®, Rebif® or Extavia®) + oral daily placebo
  Arms: GA or IFN + Placebo

SUMMARY:
A multinational, multicenter, randomized, double-blind, parallel-group, placebo-controlled study to assess the safety, tolerability and efficacy of two daily doses of oral laquinimod (0.6mg or 1.2mg) in adjunct to glatiramer acetate (GA) or interferon-beta (IFN-B) in relapsing remitting multiple sclerosis (RRMS) subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a documented MS diagnosis as defined by the Revised McDonald criteria [Ann Neurol 2011: 69:292-302], with a relapsing-remitting disease course.
2. Subjects must be ambulatory with an EDSS score of 1-5.5 (inclusive) at the baseline visit.
3. Subjects must be relapse-free and in a stable neurological condition and free of corticosteroid treatment [intravenous (IV), intramuscular (IM) and/or oral] 30 days prior to screening (month -1).
4. Subjects must be treated with either Copaxone® or an IFN-B preparation (Avonex®, Betaseron®/Betaferon®, Rebif® or Extavia®), at a stable dose for at least 6 months prior to the screening visit (switching between IFN-B preparations during the 6 months prior to screening is allowed; switching between any IFN-B preparation and GA, or vice versa, is exclusionary).
5. Subjects must have had experienced at least one documented relapse in the 36 weeks prior to randomization, with an incomplete recovery of the neurological functions as compared to pre-relapse status.
6. Subjects must be between 18 and 55 years of age, inclusive.
7. Women of child-bearing potential must practice an acceptable method of birth control [acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive or double-barrier method (condom or diaphragm with spermicide)].
8. Subjects must be able to sign and date a written informed consent prior to entering the study.
9. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

1. An onset of a relapse between Month -1 (Screening) and 0 (Baseline), unstable neurological condition or any treatment with corticosteroids [intravenous (IV), intramuscular (IM) and/or oral] or Adrenocorticotropic hormone.
2. Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to Screening.
3. Use of immunosuppressive including Mitoxantrone (Novantrone®) or cytotoxic agents within 6 months prior to the screening visit.
4. Previous use of either of the following: natalizumab (Tysabri®), cladribine, laquinimod, and fingolimod (Gilenya®).
5. Previous treatment with intravenous immunoglobulin (IVIG) within 2 months prior to screening visit.
6. Systemic corticosteroid treatment of ≥30 consecutive days duration within 2 months prior to screening visit.
7. Previous total body irradiation or total lymphoid irradiation.
8. Previous stem cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
9. Use of moderate/strong inhibitors of cytochrome P450 CYP3A4 within 2 weeks prior to the screening visit.
10. Use of inducers of CYP3A4 within 2 weeks prior to the screening visit.
11. Use of amiodarone within 2 years prior to screening visit.
12. Pregnancy or breastfeeding.
13. A ≥3xULN serum elevation of either alanine transaminase (ALT) or aspartate transaminase (AST) at screening.
14. Serum direct bilirubin which is ≥2x upper limit of normal (ULN) at screening.
15. Subjects with a potentially clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical examinations, ECG, laboratory tests or chest X-ray. Such conditions may include (but are not limited to):

    * A cardiovascular or pulmonary disorder that cannot be well-controlled by standard treatment permitted by the study protocol.
    * A gastrointestinal disorder that may affect the absorption of study medication.
    * Renal or metabolic diseases
    * Any form of acute or chronic liver disease
    * Known human immunodeficiency virus (HIV) positive status
    * A history of drug and/or alcohol abuse
    * An unstable psychiatric disorder.
    * A known history of tuberculosis.
    * Unstable psychiatric disorder
    * Any malignancies, excluding basal cell carcinoma (BCC), in the last 5 years.
16. A glomerular filtration rate less than 60 ml/min at screening visit.
17. A known history of sensitivity to gadolinium (Gd).
18. Inability to successfully undergo MRI scanning.
19. Previous endovascular treatment for Chronic Cerebrospinal Venous Insufficiency (CCSVI).
20. Known drug hypersensitivity that would preclude administration of laquinimod, such as hypersensitivity to: mannitol, meglumine or sodium stearyl fumarate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy | 10 months
  To assess the safety, tolerability and efficacy of laquinimod in RRMS

SECONDARY OUTCOMES:
Tolerability | 10 months
  To assess the safety, tolerability and efficacy of laquinimod in RRMS as compared to placebo, subjects treated with GA or an IFN-B preparation (Avonex®, Betaseron®/Betaferon®, Rebif® or Extavia®).

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Gold, MD, Principal Investigator